CLINICAL TRIAL: NCT05181839
Title: An Observational, Prospective, European, Multicentre, Mixed Methods Study to Describe the Lived Experience of X-Linked Hypophosphatemia (XLH) for Adolescents at End of Skeletal Growth
Brief Title: A Study to Describe the Lived Experience of XLH for Adolescents at End of Skeletal Growth
Status: Completed | Type: Observational
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: 2020-70-EU-CRY
Record Dates: First submitted 2021-11-15; First posted 2022-01-06 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: X-Linked Hypophosphatemia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Burosumab — To describe the lived experience of XLH for adolescents who are being treated with burosumab at the end of skeletal growth with a focus on adolescent-reported symptoms, activity duration and intensity, and wider burden, describing change over time for those who continue and discontinue burosumab after the end of skeletal growth.

SUMMARY:
An observational, prospective, mixed-methods study involving the integration of quantitative and qualitative data exploring the lived experience of burosumab-treated adolescents with XLH at the end of skeletal growth.

DETAILED DESCRIPTION:
This an observational, prospective, European, multicentre, mixed methods study that will involve the integration of quantitative and qualitative data exploring the lived experience of burosumab-treated adolescents with XLH at the end of skeletal growth. The study will involve two observation periods around the confirmed date of end of skeletal growth (index date)

The purpose of this study is to describe the lived experience of XLH for adolescents who are being treated with burosumab at the end of skeletal growth, with a focus on adolescent reported symptoms, activity duration and intensity, and wider burden, and to describe change over time for those who continue and discontinue burosumab at the end of skeletal growth. The study will also explore the experiences of carers at the time the adolescent reaches the end of skeletal growth.

The key objectives of this study are to:

1. Describe the lived experience of adolescents with XLH who are being treated with burosumab within the 12 weeks prior to reaching the end of skeletal growth.
2. Describe the lived experience of adolescents with XLH during the 26 weeks immediately after the end of skeletal growth, overall and according to whether they continue or discontinue burosumab treatment.
3. Describe within-person changes in the lived experience of adolescents with XLH after reaching end of skeletal growth, in relation to their own pre-end of skeletal growth period.
4. Explore the supportive care needs and burden on carers at the time the adolescent with XLH reaches end of skeletal growth.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of XLH (documented diagnosis of XLH in medical records, and evidence of at least one of the following: hypophosphataemia and/or impaired phosphate reabsorption due to elevated FGF23; PHEX mutation).
* Aged 12 to 17 years at start of study.
* Has open growth plates at enrolment and is estimated by their treating clinician to reach end of skeletal growth within the next 26 weeks (based on clinician's judgement in accordance with their normal approach used in routine practice).
* Has been receiving treatment with burosumab for at least study le (52 weeks).
* Provides informed consent to take part in the study (or provides assent, and carer provides consent, where applicable in accordance with specific country regulations).

Carer Inclusion Criteria:

* A main carer of a study participant (i.e. a parent or guardian who provides day-today support or care for the adolescent with XLH who is taking part in this study).
* Provides informed consent to take part in the study (for self and/or on behalf of eligible adolescent, where applicable in accordance with specific country regulations).

Exclusion Criteria:

* Unwilling and unable to participate in all aspects of the study (i.e. interviews, app, EQ- 5D-Y, wearable data collection) and /or does not agree to the collection of data from medical records.
* Missed two or more injections of burosumab in the past 6 months.
* Is planned to have any surgery during the study period.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population for this study is adolescents with XLH approaching end of skeletal growth, who are being treated with burosumab for at least 12 months as part of routine clinical care at specialist paediatric centres within the UK, France, Germany, Spain and the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Describe the lived experience of adolescents with XLH who are being treated with burosumab within the 12 weeks prior to reaching the end of skeletal growth. | 12 Weeks
Describe the lived experience of adolescents with XLH during the 26 weeks immediately after the end of skeletal growth, overall and according to whether they continue or discontinue burosumab treatment. | 26 weeks
Describe within-person changes in the lived experience of adolescents with XLH after reaching end of skeletal growth, in relation to their own pre-end of skeletal growth period. | Up to 52 weeks
Explore the supportive care needs and burden on carers at the time the adolescent with XLH reaches end of skeletal growth. | will be completed between weeks 21 and 25

CONTACTS AND LOCATIONS:
Locations (14):
- France (3):
  - Centre Hospitalier Universitair de Lille, Lille
  - Hospices Civils De Lyon, Lyon
  - APHP Paris - Assistance Publique Hopitaux de Paris, Paris
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- University Medical Center Groningen - Beatrix Children's Hospital, Groningen, Netherlands
- Spain (4):
  - Hospital Saint Joan de Deu, Barcelona, Catalona
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Universitario Virgen a de las Nieves, Granada
- United Kingdom (5):
  - Royal Manchester Childrens Hospital, Manchester, Greater Manchester
  - Birmingham Women's and Children's Hospital, Birmingham
  - Bristol Royal, Bristol
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: No